CLINICAL TRIAL: NCT04920461
Title: Visual-spatial and Visual-perceptual Disorders Following Cerebellar Strokes
Acronym: VISUO-CEREBRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2019/423
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Stroke, Ischemic; Cerebellar Lesions
MeSH Terms: conditions — Ischemic Stroke | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Additional MRI sequences (Experimental)
  Interventions: Device: Additional MRI sequences; Other: Neuropsychological assessment

INTERVENTIONS:
Device: Additional MRI sequences — Additional MRI sequences (3D T2 SPACE sequence, 4/5 minutes approximatively)
Other: Neuropsychological assessment — Neurovisual function assessed with neuropsychological tests

SUMMARY:
This study aims at assessing the proportion of patients suffering from neuro-visual troubles (visual-spatial and/or visual-perceptual ), after cerebellar strokes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Being able to pass initial neuropsychological tests within 10 days after stroke

Exclusion Criteria:

* Previous central neural system/psychiatric/eye disease (including severe cranial trauma)
* Chronic alcoholism
* MRI contraindication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Presence of Neuro-Visual Disorder | Month 3
  Presence of neuro-visual disorder will be confirmed by obtaining at least 2 pathological scores at following neuropsychological tests:
  * Rey & Taylor figures (score from 0 to 36, maximum)
  * Judgment of Line Orientation (score from 0 to 36, maximum)
  * Weschler Adult Intelligence Scale (final score is intelligence quotient, with an average score is fixed at 100)
  * Test of Attentional Performance
  * Visual Object and Space Perception Battery (eight tests each designed to assess a particular aspect of object or space perception, while minimising the involvement of other cognitive skills)
  * Visual agnosia assesment protocole (noted on 10 points)

CONTACTS AND LOCATIONS:
Overall Officials: Eloi MAGNIN, MD, PhD, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No